CLINICAL TRIAL: NCT02288052
Title: Consolidation of Motor Learning of Writing Skills and Its Related Brain Activity Changes in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Alice Nieuwboer, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: G.0906.11
Record Dates: First submitted 2014-11-03; First posted 2014-11-11 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson Disease
Keywords: Handwriting; Motor learning
MeSH Terms: conditions — Parkinson Disease | interventions — Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Writing program (Experimental): The program will train participants in maintaining writing amplitude, writing speed, writing fluently and automatization of writing.
  Interventions: Behavioral: Writing program
- Stretch & Relaxation program (Placebo Comparator): The program will learn participants to alleviate tension in the upper limbs and will consist of exercises performed while lying down or sitting.
  Interventions: Behavioral: Stretch & Relaxation program

INTERVENTIONS:
Behavioral: Writing program — 6 weeks of at-home training (5days/week, 30minutes/day) using both pen-and-paper exercises and exercises on a writing tablet.
  Arms: Writing program
Behavioral: Stretch & Relaxation program — 6 weeks of at-home training (5days/week, 30minutes/day) using a DVD with exercises.
  Arms: Stretch & Relaxation program

SUMMARY:
The basal ganglia play an important role in motor learning, especially during the consolidation phase of motor learning. This raises the question whether it is possible to sustain learning increments in a neurodegenerative condition such as Parkinson's disease (PD). The aim of this study is to gain knowledge on whether it is possible to relearn skills which are actually affected by PD, such as writing, and determine whether neuroplasticity is possible. In this randomized controlled study, PD patients will either follow intensive writing training or a placebo treatment (stretch and relaxation training) during 6 weeks. The writing training will focus on automatization (withstanding dual task interference), transfer to an untrained task and retention. The placebo program is aimed to reduce stiffness in the upper limbs and has been shown to be ineffective in PD. To date, it is unknown how neural networks change as a result of consolidation after a prolonged period of motor learning in PD. Therefore the second arm of this study will investigate, for the first time, changes in neural connectivity using brain imaging data to elucidate which neuroanatomical regions are involved in consolidation of learning in PD. Finally, DTI and resting state fMRI-analysis will complement insights into the neural changes as a result of learning.

DETAILED DESCRIPTION:
This translational study is a monocentric Randomized Controlled Trial (RCT). The investigators will recruit 40 PD patients from the early Hoehn & Yahr stages. Patients will be randomly allocated to an experimental group (writing training) and a control group (stretch- and relaxation training). All patients will receive the same frequency and duration of intervention. After the training period, patients will be followed up for another 6 weeks. Patients will be tested in the ON-phase of the medication cycle at 3 occasions: before (T1) and after training (T2) and after a 6-week retention period (T3). At T1 & T2 participants will be tested at the behavioral & neural level. At T3 participants will only be tested at the behavioral level.

Motor performance will be measured using MRI-compatible touch sensitive tablets and pencils. This system allows registration and translation of writing movements into online-cursor movements on screen in and outside a scanner environment. Both patient groups will be compared during a behavioral test battery consisting of (i) a trained sequence with and without visual cues; (ii) an untrained sequence with and without visual cues to test transfer; and (iii) a trained dual task to test automatization. Visual cues will consist of differently colored target zones of different band widths, indicating the scale and accuracy of writing.

Functional MRI measurements will take place in a 3T MR Philips Intera scanner. Before scanning, subjects will undergo a training session in a dummy scanner to familiarize them with the scanner environment and task instructions. During the fMRI sessions, participants will perform a trained and untrained sequence, both with and without visual cues. To control for differences in movement speed, all participants will perform the tasks at the same frequency, defined by an auditory pace. In addition to the fMRI measurements, resting state fMRI and DTI will also be performed to reveal alterations of the structural and functional connectivity between critical regions.

Behavioral data will be recorded as xy-coordinates and pressure values at a sampling rate of 200Hz and with a spatial resolution of 32.5µm. Statistical analysis of the behavioral data will have a between-subject factor of group (experimental and placebo group) and a within-subject factor of time (before training, after training and after the retention period).

Image analysis will be performed with Statistical Parametric Mapping (SPM) software. The investigators will contrast for either decreased or increased activation, as different regions may show divergent changes related to learning and transfer, with group as a between-subject factor and time (before and after training) and task condition (trained with cues, trained without cues, untrained with cues and untrained without cues) as within-subject factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD based on the UK Brain Bank criteria
* Hoehn & Yahr stage I (with impairments on the right side) and II in the on-phase
* Without cognitive impairment (MMSE >24)
* On stable medication
* Right handed

Exclusion Criteria:

* Deep Brain Stimulator
* Other contra-indications for MR scanning
* Colorblind

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in writing amplitude (cm) on tablet after 6 weeks of training | 6 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Change from baseline in writing amplitude (cm) on tablet after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Change from baseline in brain activity during writing (functional MRI) after 6 weeks of training | 6 weeks
  Analysis of the change in Blood Oxygen Level Dependent (BOLD) response
Change from baseline in brain activity during rest (resting state MRI) after 6 weeks of training | 6 weeks
  Analysis of the change in Blood Oxygen Level Dependent (BOLD) response
Change from baseline in Diffusion Tensor Imaging after 6 weeks of training | 6 weeks
  Analysis of the change in Blood Oxygen Level Dependent (BOLD) response

SECONDARY OUTCOMES:
Transfer of change in writing amplitude to an untrained writing sequence after 6 weeks of training | 6 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Transfer of change in writing amplitude to an untrained writing sequence after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Change from baseline in dual task effect (DTE) for writing amplitude after 6 weeks of training | 6 weeks
  Analysis of the DTE using the following formula: DTE= ((dual task amplitude-single task amplitude)/(single task amplitude))*100
Change from baseline in dual task effect (DTE) for writing amplitude after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis of the DTE using the following formula: DTE= ((dual task amplitude-single task amplitude)/(single task amplitude))*100
Change from baseline in writing fluency (normalized jerk) on tablet after 6 weeks of training | 6 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Change from baseline in writing fluency (normalized jerk) on tablet after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis based on measurement of XYZ coordinates, measured at a spatial resolution of 32.5 μm.
Systematic Screening of handwriting difficulties (writing on paper) - change from baseline in quality score after 6 weeks of training | 6 weeks
  Analysis of the quality of handwriting based on different criteria (fluency in letter formation, connections between letters, regularity of letter height, space between words and straightness of the sentence).
Systematic Screening of handwriting difficulties (writing on paper) - change from baseline in quality score after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis of the quality of handwriting based on different criteria (fluency in letter formation, connections between letters, regularity of letter height, space between words and straightness of the sentence).
Systematic Screening of handwriting difficulties (writing on paper) - change from baseline in writing speed after 6 weeks of training | 6 weeks
  Analysis of the number of letters written within a period of 5 minutes.
Systematic Screening of handwriting difficulties (writing on paper) - change from baseline in writing speed after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis of the number of letters written within a period of 5 minutes.
Change from baseline in Purdue Pegboard test after 6 weeks of training | 6 weeks
  Analysis of the number of pegs placed within 30s.
Change from baseline in Purdue Pegboard test after 12 weeks, including 6 weeks without training | 12 weeks
  Analysis of the number of pegs placed within 30s.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Nieuwboer, Professor, Principal Investigator — KU Leuven
Locations (1):
- Department of Rehabilitation Sciences KU Leuven, Leuven, Belgium

REFERENCES:
- [Background] Broeder S, Nackaerts E, Nieuwboer A, Smits-Engelsman BC, Swinnen SP, Heremans E. The effects of dual tasking on handwriting in patients with Parkinson's disease. Neuroscience. 2014 Mar 28;263:193-202. doi: 10.1016/j.neuroscience.2014.01.019. Epub 2014 Jan 19. PMID 24447597
- [Background] Nackaerts E, Vervoort G, Heremans E, Smits-Engelsman BC, Swinnen SP, Nieuwboer A. Relearning of writing skills in Parkinson's disease: a literature review on influential factors and optimal strategies. Neurosci Biobehav Rev. 2013 Mar;37(3):349-57. doi: 10.1016/j.neubiorev.2013.01.015. Epub 2013 Jan 16. PMID 23333265
- See also: Neuromotor Rehabilitation Research Group KU Leuven — https://gbiomed.kuleuven.be/english/research/50000743/nrrg1/nrrg.htm